CLINICAL TRIAL: NCT01942122
Title: Role of DLBS1442 for The Treatment of Pain in Patients Suspected Endometriosis
Brief Title: DLBS1442 for The Treatment of Pain in Patients Suspected Endometriosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dexa Medica Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DLBS1442-0212
Record Dates: First submitted 2013-09-10; First posted 2013-09-13 (Estimated); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Endometrioma; Visual Analogue Pain Scale: Moderate or Severe Pain
Keywords: DLBS1442; Endometriosis; Pain; Visual Analogue Scale; Endometriosis Health Profile (EHP-30TM)
MeSH Terms: conditions — Endometriosis; Pain | interventions — Mefenamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- DLBS1442 100 (Experimental): DLBS1442 capsules 3x100 mg daily, taken every day along the study period
  Interventions: Drug: DLBS1442 100
- DLBS1442 200 (Experimental): DLBS1442 capsules 3x200 mg daily, taken every day along the study period
  Interventions: Drug: DLBS1442 200
- Mefenamic acid (Active Comparator): Mefenamic acid tablets 3 x 500 mg daily, only taken for five (5) days during the menstrual period, i.e. day 1st to day 5th of menstrual period.
  Interventions: Drug: Mefenamic acid

INTERVENTIONS:
Drug: DLBS1442 100 — Study treatment will be DLBS1442 capsules at a dose of 3x100 mg daily. DLBS1442 will be taken every day for 8 weeks (2 menstrual cycles).
  Other Names: Dismeno 100
  Arms: DLBS1442 100
Drug: Mefenamic acid — Control will be mefenamic acid 500 mg tablets, administered 3 times daily for 5 days during the menstrual period, i.e. day 1st to day 5th of the menstrual period. The drug will be given within the 8 weeks of study period (2 menstrual cycles).
  Other Names: Pondex Forte
  Arms: Mefenamic acid
Drug: DLBS1442 200 — Study treatment will be DLBS1442 capsules at a dose of 3x200 mg daily. DLBS1442 will be taken every day for 8 weeks (2 menstrual cycles).
  Other Names: Dismeno 200
  Arms: DLBS1442 200

SUMMARY:
This is a 3-arm, prospective, randomized, double-blind, and controlled study of DLBS1442 for the treatment of pain in patients suspected endometriosis. It is hypothesized that the reduction of the composite-pain intensity (as measured by VAS) from baseline to the end of study (week 8th) resulting from administration of DLBS1442, regardless of the dosage regimen, is significantly greater than that of Control. In addition, the administration of DLBS1442 at higher dose also results in significantly greater reduction than that of DLBS1442 at lower dose and of Control.

DETAILED DESCRIPTION:
There will be three groups of treatment by dosage regimen in this study. Eligible subjects will be randomized to receive any of the following regimens: 1) DLBS1442 at a dose of 3 x 100 mg daily, or 2) DLBS1442 at a dose of 3 x 200 mg daily; or 3) mefenamic acid at a dose of 3 x 500 mg daily. DLBS1442 will be taken every day along the study period (8 weeks), while mefenamic acid will only be taken for five (5) days during the menstrual period, i.e. day 1st to day 5th of menstrual period. Study treatment will be given at a standardized starting point for all subjects, i.e. on the first day of their respective menstrual periods. Clinical and laboratory examinations to evaluate the investigational drug's efficacy and safety will be performed at baseline and every 4-week interval throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent before any trial related activities
* Female of 18 - 50 years of age
* Subjects suspected with cystic endometriosis or adenomyosis confirmed by transvaginal ultrasonography (or transrectal ultrasonography for unmarried subjects)
* Presence of moderate or severe pain as shown by VAS score of at least 4 on at least one of the following pain: menstrual pain (dysmenorrhea), dyspareunia, non-menstrual pelvic pain, dysuria, dyschezia
* Occurrence of at least 3 last sequential menstrual cycles of 21 - 35 days duration prior to screening

Exclusion Criteria:

* Pregnancy
* Patients with infertility who are willing to be pregnant
* Using hormonal contraception or other forms of hormonal therapy within the last 30 days
* Being under therapy with systemic corticosteroids on a chronic or regular basis within the last 90 days
* History or presence of suspected malignancy abnormalities
* History of surgical treatment for endometriosis within 3 months prior to screening
* History of hysterectomy or oophorectomy
* Presence of clinical signs of sexually transmitted disease
* Presence of unexplained uterine or cervical bleeding
* Impaired liver function: serum ALT > 2.5 times upper limit of normal
* Impaired renal function: serum creatinine >= 1.5 times upper limit of normal
* Known or suspected allergy to similar products

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-10; Primary Completion 2021-02 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
Reduction of intensity (VAS) of composite-pain | Week 8
  Reduction of the intensity of composite-pain (dysmenorrhea, dyspareunia, non-menstrual chronic pelvic pain, dysuria, dyschezia) as measured by Visual Analogue Scale (VAS).

SECONDARY OUTCOMES:
Reduction of the intensity of each pain (VAS) | Week 4, week 8
  Reduction of the intensity of each pain (dysmenorrhea, dyspareunia, non-menstrual chronic pelvic pain, dysuria, dyschezia) as measured by Visual Analogue Scale (VAS).
Response rate | Week 8
  Response rate is defined as percentage of subjects at the end of study experiencing a reduction of VAS score of >= 3 or >= 30% as compared to baseline, in each of the composite pain found at baseline (i.e. dysmenorrhea, dyspareunia, non-menstrual pelvic pain, dysuria, or dyschezia).
Improvement of quality of life | Week 4, week 8
  Improvement of quality of life is measured by Endometriosis Health Profile (EHP-30) questionnaire score.
Serum CA-125 | Week 8
  Reduction in serum CA-125 level.
IL-6 | Week 8
  Change of IL-6
Number of rescue medication | During the course of the study
  Number of rescue medication (pain relieving drug, i.e. ibuprofen 400 mg tablet) needed during the course of the study.
Pain-free period | During the course of the study
  Time to the first day on which subjects take rescue medication.
Percentage or proportion of subjects who complete the study | Week 8
  Percentage or proportion of subjects who complete the study (2 cycles).
ECG | Week 8
  Electrocardiography.
Vital signs | Week 4, week 8
  Vital signs measured include: blood pressure, heart rate, respiratory rate.
Liver function | Week 8
  Liver function measured includes: serum ALT (SGPT), serum AST (SGOT), and alkaline phosphatase (AP).
Renal function | Week 8
  Renal function measured includes: serum creatinine and blood urea nitrogen (BUN).
Routine hematology | Week 8
  Routine hematology measured includes: hemoglobin, hematocrit, RBC, WBC, differentiation of WBC, and platelet count.
Adverse event | During the course of the study
  Adverse event will be observed and managed along the study course.
Reduction of intensity (VAS) of composite-pain | 4 weeks
  Reduction of the intensity of composite-pain (dysmenorrhea, dyspareunia, non-menstrual chronic pelvic pain, dysuria, dyschezia) as measured by Visual Analogue Scale (VAS).
hs-CRP | Week 8
  Change in serum hs-CRP.

CONTACTS AND LOCATIONS:
Overall Officials: Kanadi Sumapraja, SpOG(K), MD, Principal Investigator — Division of Reproductive, Endocrinology, and Infertility, Department of Obstetrics and Gynecology, Faculty of Medicine, University of Indonesia/Dr. Cipto Mangunkusumo Hospital
Locations (3):
- Indonesia (3):
  - Yasmin Clinic, Dr. Cipto Mangunkusumo Hospital (Kencana), Jakarta Pusat, Jakarta Special Capital Region
  - Department of Obstetrics and Gynecology, RSUP Persahabatan, Jakarta Pusat, Jakarta Special Capital Region
  - Department of Obstetrics and Gynecology RSUP Fatmawati, Jakarta